CLINICAL TRIAL: NCT07363759
Title: ISOVUE Contrast for Intraoperative Assessment of Discectomy Quality in TLIF: A Prospective Randomized Trial
Brief Title: ISOVUE Comparative Trial
Acronym: ISOVUE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rush University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 18072502-IRB02
Record Dates: First submitted 2026-01-07; First posted 2026-01-23 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Lumbar Degenerative Disease; Lumbar Degenerative Disc Disease; Degenerative Spine
Keywords: isovue; iodinated contrast
MeSH Terms: conditions — Intervertebral Disc Degeneration

STUDY DESIGN:
Intervention Model Description: After obtaining informed consent, patients were randomized into either a control (Observation) or investigational (Feedback) group. In the observation group, after initial discectomy, ISOVUE M300 contrast was administered into the disc space via angiocatheter to assess the extent of discectomy by obtaining orthogonal radiographs of the contrast-enhanced space. Then, the contrast agent was extracted via suction and the disc space was irrigated with saline. The case then proceeded with graft/cage insertion without additional excision. In the feedback group, prior to graft/cage insertion, the surgeon used the contrast feedback to enhance the preparation.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Observation (Placebo Comparator): In the Observation group, after initial discectomy and endplate preparation, ISOVUE-300M contrast was administered into the disc space and orthogonal anterior-posterior and lateral radiographs were obtained. The case then proceeded with graft and cage insertion without additional disc excision or endplate work.
  Interventions: Procedure: ISOVUE 300 Observation
- Feedback (Experimental): In the Feedback group, the surgeon was permitted to utilize the ISOVUE imaging as a feedback mechanism to then re-prepare the disc space prior to final graft/cage insertion. An additional dose of ISOVUE-300M was administered into the disc space with repeat radiographs obtained prior to grafting/cage insertion to demonstrate the effect of the second pass of disc and cartilage removal.
  Interventions: Procedure: ISOVUE 300 Feedback

INTERVENTIONS:
Procedure: ISOVUE 300 Observation — In the Observation group, after initial discectomy and endplate preparation,ISOVUE-300M contrast was administered into the disc space and orthogonal anterior-posterior and lateral radiographs were obtained. The case then proceeded with graft and cage insertion without additional disc excision or endplate work.
  Arms: Observation
Procedure: ISOVUE 300 Feedback — In the Feedback group, the surgeon was permitted to utilize the ISOVUE imaging as a feedback mechanism to then re-prepare the disc space prior to final graft/cage insertion. An additional dose of ISOVUE-300M was administered into the disc space with repeat radiographs obtained prior to grafting/cage insertion to demonstrate the effect of the second pass of disc and cartilage removal.
  Arms: Feedback

SUMMARY:
This study aimed to investigate a novel technique for intraoperative quantitative and qualitative feedback during discectomy and endplate preparation in TLIF.

DETAILED DESCRIPTION:
The purpose of this study was to introduce a novel surgical technique using ISOVUE-300M contrast dye for intraoperative visualization of discectomy progress and to test the value of this technique by comparing outcomes of two patient cohorts. The investigators hypothesize that the standard TLIF technique results in a surprisingly low percentage of effective disc preparation, even when performed by an experienced TLIF surgeon. Secondly, the investigators hypothesize that by using intraoperative visual feedback to guide a second discectomy pass that the extent of disc space preparation can be substantially improved compared to patients where visual feedback is not available. Lastly, the investigators aim to conduct a clinical outcomes analysis evaluating radiographic and complication outcomes. To the best of the authors' knowledge, this prospective study is the first to evaluate differences in disc space preparation using a novel contrast-based technique while also providing clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing open circumferential transforaminal lumbar interbody fusion or midline cortical TLIF for degenerative spondylolisthesis

Exclusion Criteria:

* All not in the group above

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2019-04-11 (Actual); Primary Completion 2023-06-19 (Actual); Study Completion 2023-06-19 (Actual)

PRIMARY OUTCOMES:
Anteroposterior Plane Clearance | Immediately after Discectomy
  Disc space clearance in the anteroposterior (AP) plane at the index level measured on oblique radiographs.
Mediolateral Plane Clearance | Immediately after Discectomy/Excision Intraoperatively
  Disc space clearance in the mediolateral (ML) plane as measured by oblique radiographs.
Visual Analog Scale | First Postoperative Clinic Appointment (within first 6 weeks)
  Visual Analog Scale survey assessing leg pain and back pain

SECONDARY OUTCOMES:
Lumbar Lordosis | Immediately after Discectomy Intraoperatively
  Lumbar Lordosis as measured by oblique radiographs.
Pelvic Incidence | Immediately after Discectomy Intraoperatively
  Pelvic incidence (PI) as measured by oblique radiographs.
Disc Height | Immediately after Discectomy Intraoperatively
  Disc height at the index level as identified by oblique radiographs.
Oswestry Disability Index | First Postoperative Clinic Appointment (within first 6 weeks)
  Oswestry Disability Index survey describing disability as a result of spinal conditions.
Short Form Survey | First Postoperative Clinic Appointment (within first 6 weeks)
  SF-12 survey asking patient views about health

CONTACTS AND LOCATIONS:
Locations (1):
- Rush University Medical Center, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No
The investigators will consider sharing if contacted with reasonable requests.

REFERENCES:
- [Background] de Kunder SL, van Kuijk SMJ, Rijkers K, Caelers IJMH, van Hemert WLW, de Bie RA, van Santbrink H. Transforaminal lumbar interbody fusion (TLIF) versus posterior lumbar interbody fusion (PLIF) in lumbar spondylolisthesis: a systematic review and meta-analysis. Spine J. 2017 Nov;17(11):1712-1721. doi: 10.1016/j.spinee.2017.06.018. Epub 2017 Jun 21. PMID 28647584
- [Background] Lan T, Hu SY, Zhang YT, Zheng YC, Zhang R, Shen Z, Yang XJ. Comparison Between Posterior Lumbar Interbody Fusion and Transforaminal Lumbar Interbody Fusion for the Treatment of Lumbar Degenerative Diseases: A Systematic Review and Meta-Analysis. World Neurosurg. 2018 Apr;112:86-93. doi: 10.1016/j.wneu.2018.01.021. Epub 2018 Jan 31. PMID 29367001
- [Background] Katuch V, Grega R, Knorovsky K, Banoci J, Katuchova J, Sasala M, Ivankova H, Kapralova P. Comparison between posterior lumbar interbody fusion and transforaminal lumbar interbody fusion in the management of lumbar spondylolisthesis. Bratisl Lek Listy. 2021;122(9):653-656. doi: 10.4149/BLL_2021_105. PMID 34463112
- [Background] Reitman CA, Anderson DG, Fischgrund J. Surgery for degenerative spondylolisthesis: open versus minimally invasive surgery. Clin Orthop Relat Res. 2013 Oct;471(10):3082-7. doi: 10.1007/s11999-013-3171-8. Epub 2013 Jul 20. No abstract available. PMID 23873608